CLINICAL TRIAL: NCT04229537
Title: To Evaluate Safety and Efficacy of SCT-I10A Combined SCT200 or SCT-I10A Combined SCT200 Plus Chemotherapy in Advanced Esophageal Squamous Cell Carcinoma and Colorectal Cancer: a Phase Ⅰb, Open-label, Multicenter Study
Brief Title: Study of SCT-I10A Combined SCT200 or SCT-I10A Combined SCT200 Plus Chemotherapy in ESCC and CRC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT-I10A-X102
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Colorectal Cancer
Keywords: SCT-I10A; SCT200
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCT-I10A combined SCT200 in ESCC (Experimental): SCT-I10A: 200 mg intravenous (IV) on Day 1 of Q3W. SCT200: 6mg/kg intravenous (IV) on Day 1 of QW, then 8mg/kg intravenous (IV) on Day 1 of Q2W
  Interventions: Biological: SCT-I10A; Biological: SCT200
- SCT-I10A combined SCT200 in CRC (Experimental): SCT-I10A: 200 mg intravenous (IV) on Day 1 of Q3W. SCT200: 6mg/kg intravenous (IV) on Day 1 of QW, then 8mg/kg intravenous (IV) on Day 1 of Q2W
  Interventions: Biological: SCT-I10A; Biological: SCT200
- SCT-I10A combined SCT200 plus Chemotherapy in CRC (Experimental): SCT-I10A: 200 mg intravenous (IV) on Day 1 of Q3W. SCT200: 6mg/kg intravenous (IV) on Day 1 of QW, then 8mg/kg intravenous (IV) on Day 1 of Q2W.
  Chemotherapy: Capecitabine and Oxaliplatin.
  Interventions: Biological: SCT-I10A; Biological: SCT200; Other: Chemotherapy

INTERVENTIONS:
Biological: SCT-I10A — 200 mg intravenous (IV) on Day 1 of Q3W.
Biological: SCT200 — 6mg/kg intravenous (IV) on Day 1 of QW, then 8mg/kg intravenous (IV) on Day 1 of Q2W
Other: Chemotherapy — Capecitabine and Oxaliplatin.
  Arms: SCT-I10A combined SCT200 plus Chemotherapy in CRC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SCT-I10A combined SCT200 or SCT-I10A combined SCT200 plus chemotherapy in advanced esophageal squamous cell carcinoma and colorectal cancer

DETAILED DESCRIPTION:
This is a open label, multicenter, phase III study designed to evaluate the safety and efficacy in advanced esophageal squamous cell carcinoma and colorectal cancer treated with SCT-I10A combined SCT200 or SCT-I10A combined SCT200 plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent before screening；
* Males or females. Aged 18 to 75 years old;
* Life expectancy≥12 weeks before starting treatment (clinical assessment);
* With an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* Histologically or cytologically confirmed advanced esophageal squamous cell carcinoma or colorectal cancer;
* Patients with advanced esophageal squamous cell carcinoma undergoing first-line systemic chemotherapy progression or intolerance were included in Arm 1; Patients with RAS and BRAF wild-type advanced colorectal cancer undergoing at least second line systemic chemotherapy progression or intolerance were included in Arm 2; Patients with RAS and BRAF wild-type advanced colorectal cancer untreated with cetuximab were included in Arm 3;
* According to RECIST 1.1, patients must have at least one measurable lesion that can be accurately assessed;
* Adequate organ and bone marrow function as defined below:

Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 100×109/L; Hemoglobin greater than/equal to 90g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 3 times ULN, or less than/equal to 5 times ULN if known liver metastases; Total bilirubin less than/equal to 1.5 times ULN; Serum creatinine less than/equal to 1.5 times ULN or Ccr>60ml/min; Thyroid stimulating hormone (TSH) hormone levels less than/equal to ULN; Serum magnesium greater than/equal to ULN; APTT, INR, PT less than/equal to 1.5 times ULN.

Exclusion Criteria:

* Patients who were allergic to analogue of SCT-I10A/SCT200 and/or its inactive ingredients, Patients who were allergic to Capecitabine and/or Oxaliplatin were also excluded in cohort3;
* Patients have been treated with anti-PD-L1/PD-L2 or anti-PD-1, EGFR antibody or EGFR-TKI;
* Within 4 weeks prior to the first dose of study drug, patients have received anti-tumor drugs (such as chemotherapy, endocrine therapy, targeted therapy, immune therapy, tumor embolization). Within 6 weeks prior to the first dose of study drug, patients have been treated with biological products, nitrosourea or mitomycin C. Within 4 weeks prior to the first dose of study drug, patients have been treated with tumor embolization or radiotherapy;
* Within 2 weeks prior to the first dose of study drug, patients have received corticosteroids or other immunosuppressive agents;
* Within 1 month prior to the first dose of study drug, patients have received live attenuated vaccine (LAV);
* Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices;
* Patients with significant malnutrition. Patients will be excluded if they are receiving intravenous hyperalimentation, or require continuous infusion therapy with hospitalization. Patients whose nutrition has been well controlled for ≥ 28 days prior to randomization may be enrolled.
* Within 4 weeks prior to the first dose of study drug, patients have received major surgery, or had wounds, ulcers or fractures that haven't healed; Within 6 weeks prior to the first dose of study drug, patients were suffering with gastrointestinal perforation or fistula;
* Has active infection or fever of unknown origin(> 38.5℃)；
* Has invaded large vessels and weasand
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previous treated brain metastases may participate provided they are stable for at least 2 weeks prior to the first dose of study medication, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. Subjects with asymptomatic brain metastases (without neurological symptoms, not using steroids, tumor lesions≤1.5cm) may participate in condition that the tumor lesion should be regularly evaluated using identical imaging modality for each assessment, either MRI or CT scans;
* Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
* Poorly controlled hypetension. Within 6 months prior to study, patients had uncontrolled concurrent diseases, including but not limited to acute myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack, congestive heart failure (NYHA, greater than II), left ventricular ejection fraction (LVEF) <50%, and with related heart disease.
* Patients who have interstitial lung disease or imaging features of interstitial pneumonia, or who have history of non-infectious pneumonia treated with corticosteroids.
* Patients with an active, known or suspected autoimmune disease or a history of autoimmune disease;
* Within 5 year prior to the first dose of study drug, patients have other primary malignancies;
* Have a history of HIV;
* Patients with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C(e.g. HCV RNA [quantitative] is detected);
* Prior to the first dose of study drug, patients had toxicity due to previous anti-tumor treatment, which hasn't return to Grade 0-1 according to the NCI CTCAE v5.0;
* Has known with alcohol or drug addiction;
* Pregnant or lactating women;
* Patients who were not willing to accept effective contraceptive measures during treatment and within 6 months after treatment;
* Subjects who are considered not suitable for the study by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 24 months
  Including adverse events and safety of laboratory tests

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 or Lugano 2014 criteria during trial treatment
Duration of response (DOR) | 24 months
  DOR is defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1 or Lugano 2014 criteria, until the date that progressive disease (PD) is objectively documented or death, whichever occurs first
Disease control rate (DCR) | 24 months
  The achievement of any a stable response（SD）, partial response (PR) or complete response (CR), according to RECIST v1.1 or Lugano 2014 criteria
Progression free survival (PFS) | 24 months
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 or Lugano 2014 criteria
Overall survival (OS) | 24 months
  OS is defined as time from first dose of SCT200 until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bai M, Lu Y, Shen L, Yin X, Gao S, Xia B, Fu Z, Zhang Z, Xie L, Ba Y. Anti-PD-1 antibody (SCT-I10A) plus anti-EGFR antibody (SCT200) in patients with advanced esophageal squamous cell carcinoma: A multicenter, open-label, phase 1b clinical trial. Cancer. 2025 Aug 15;131(16):e70046. doi: 10.1002/cncr.70046. PMID 40819238
- [Derived] Bai M, Lu Y, Shi C, Yang J, Li W, Yin X, Huang C, Shen L, Xie L, Ba Y. Phase Ib study of anti-EGFR antibody (SCT200) in combination with anti-PD-1 antibody (SCT-I10A) for patients with RAS/BRAF wild-type metastatic colorectal cancer. Cancer Biol Med. 2023 Dec 23;21(7):636-50. doi: 10.20892/j.issn.2095-3941.2023.0301. PMID 38148327